CLINICAL TRIAL: NCT01126983
Title: Lead Migration in Spinal Cord Stimulation Trials: Comparing Non-suture vs Suture and Lead Anchor Securing Methods: A Randomized Single Blind Clinical Trial for Better Outcomes.
Brief Title: Lead Migration in Spinal Cord Stimulation Trials: Comparing Non-suture vs Suture and Lead Anchor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Care, Oklahoma (Other)
Responsible Party: Spine Care of Oklahoma, Spine Care of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: spinecareleads
Record Dates: First submitted 2010-05-16; First posted 2010-05-20 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Spinal Cord Stimulation
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-Suture (Experimental): No suture will be used to secure the leads. Benzoin and Steri-Strips will be used like in the other two arms.
  Interventions: Device: Suture; Device: Lead Anchor

INTERVENTIONS:
Device: Suture — Suture (2.0 Mono-filament nylon suture) will be used to secure the leads to the skin. Benzoin and Steri-strips will also be used.
  Other Names: 2.0 Mono-filament nylon suture
Device: Lead Anchor — Suture (2.0 Mono-filament Nylon suture) will be applied over the lead anchor(Lead Anchor St.Jude Medical Co, model-long, No# 1106) to the skin. Benzion and Steri-strips will also be used.
  Other Names: 2.0 Mono-filament Nylon suture & Lead Anchor (St.Jude Medical Co) model-long, No# 1106

SUMMARY:
To assess lead migration rates using different methods of securing leads during Spinal Cord Stimulation trial period.

Spinal cord stimulation has two phases. Trial, which is a precursor for a permanent implantation. Trial lasts less than a week, which gives the patient an opportunity to assess the effectiveness of the treatment.

DETAILED DESCRIPTION:
Lead migration has been a known issue/complication with spinal cord stimulation. Lead migration during the trial period can alter the success of a trial. There is no one way of securing the leads to the skin.

Our endeavor was to look at different modes of securing the leads to the skin during the trial period and present their respective lead migration rates. The three methods are

1. suturing the leads using 2.0 mono-filament nylon to the skin,
2. suture (2.0 mono-filament nylon)over the lead anchor(St.Jude Med Co. long, model # 1106) attaching them to the skin,
3. non- suture.

In all three groups copious amounts of benzoin and steri-strips will be used.

Fluoroscopy pictures were taken after the leads were inserted and the level of the leads will be marked. After the trial period, before the leads were removed, an AP/lateral plain X-ray was taken and compared to the fluoroscopy pictures taken at the time of lead placement.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing Spinal Cord Stimulation (age > 18yrs)

Exclusion Criteria:

* patients whose trial period lasts less than 3 days or more than 5 days will be excluded from the study.
* patients that may require revision of leads or any complication that requires to take the leads out before the end of trial period.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Migration of leads with different methods of securing leads during spinal cord stimulation trial period. | 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Shadid, M.D, Principal Investigator — Spine Care of Oklahoma
Locations (1):
- Spine Care of Oklahoma, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Cameron T. Safety and efficacy of spinal cord stimulation for the treatment of chronic pain: a 20-year literature review. J Neurosurg. 2004 Mar;100(3 Suppl Spine):254-67. doi: 10.3171/spi.2004.100.3.0254. PMID 15029914
- [Background] Kemler MA, de Vet HC, Barendse GA, van den Wildenberg FA, van Kleef M. Spinal cord stimulation for chronic reflex sympathetic dystrophy--five-year follow-up. N Engl J Med. 2006 Jun 1;354(22):2394-6. doi: 10.1056/NEJMc055504. No abstract available. PMID 16738284
- [Background] Brook AL, Georgy BA, Olan WJ. Spinal cord stimulation: a basic approach. Tech Vasc Interv Radiol. 2009 Mar;12(1):64-70. doi: 10.1053/j.tvir.2009.06.007. PMID 19769908
- [Background] Holsheimer J, Barolat G, Struijk JJ, He J. Significance of the spinal cord position in spinal cord stimulation. Acta Neurochir Suppl. 1995;64:119-24. doi: 10.1007/978-3-7091-9419-5_26. PMID 8748598
- [Background] Ohnmeiss DD, Rashbaum RF. Patient satisfaction with spinal cord stimulation for predominant complaints of chronic, intractable low back pain. Spine J. 2001 Sep-Oct;1(5):358-63. doi: 10.1016/s1529-9430(01)00083-3. PMID 14588316
- [Background] Jang HD, Kim MS, Chang CH, Kim SW, Kim OL, Kim SH. Analysis of failed spinal cord stimulation trials in the treatment of intractable chronic pain. J Korean Neurosurg Soc. 2008 Feb;43(2):85-9. doi: 10.3340/jkns.2008.43.2.85. Epub 2008 Feb 20. PMID 19096610
- [Background] Rosenow JM, Stanton-Hicks M, Rezai AR, Henderson JM. Failure modes of spinal cord stimulation hardware. J Neurosurg Spine. 2006 Sep;5(3):183-90. doi: 10.3171/spi.2006.5.3.183. PMID 16961078
- [Background] Kumar K, Wilson JR, Taylor RS, Gupta S. Complications of spinal cord stimulation, suggestions to improve outcome, and financial impact. J Neurosurg Spine. 2006 Sep;5(3):191-203. doi: 10.3171/spi.2006.5.3.191. PMID 16961079
- [Background] Park CH, Huh B. Lodged spinal cord stimulator trial lead: a case report. Pain Pract. 2008 May-Jun;8(3):210-3. doi: 10.1111/j.1533-2500.2008.00199.x. PMID 18476899
- See also: Related Info — http://www.mayfieldclinic.com/PE-STIM.htm